CLINICAL TRIAL: NCT00489476
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Single Dose Efficacy and Safety Study of Staccato® Loxapine for Inhalation in Patients With Migraine Headache
Brief Title: Staccato Loxapine in Migraine (in Clinic)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexza Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMDC-104-201
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Results first posted 2017-04-24 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2008-04

CONDITIONS: Migraine
Keywords: Staccato® Loxapine, Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Loxapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 1.25 mg Staccato Loxapine (Experimental): 1.25 mg ADASUVE, single dose
  Interventions: Drug: Staccato Loxapine
- 2.5 mg Staccato Loxapine (Experimental): 2.5 mg ADASUVE, single dose
  Interventions: Drug: Staccato Loxapine
- 5 mg Staccato Loxapine (Experimental): 5 mg ADASUVE, single dose
  Interventions: Drug: Staccato Loxapine
- Staccato Placebo (Experimental): Staccato Placebo, 0 mg
  Interventions: Drug: Staccato Placebo

INTERVENTIONS:
Drug: Staccato Loxapine
  Other Names: ADASUVE
  Arms: 1.25 mg Staccato Loxapine; 2.5 mg Staccato Loxapine; 5 mg Staccato Loxapine
Drug: Staccato Placebo — Placebo aerosol inhalation (0mg)
  Arms: Staccato Placebo

SUMMARY:
The objective of this trial is to assess the efficacy and safety of Staccato Loxapine in patients with migraine headache with or without aura in a clinical setting.

DETAILED DESCRIPTION:
This study will enroll male and female patients with migraine headache with or without aura. The study will randomize ~160 patients, 1:1:1:1 to receive one of the following treatments: 1.25 mg Staccato Loxapine; 2.5 mg Staccato Loxapine; 5 mg Staccato Loxapine; Staccato Placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients between the ages of 18 to 65 years, inclusive.
2. Patients who have migraine headache with or without aura (diagnosis according to International Headache Society guidelines) for at least 6 months.
3. Patients who have a history of migraine and have had at least 3 migraine attacks in the last 3 month period (but not more than 8 migraine attacks in the last month).
4. Patients who have been pain free for at least 48 hours since the end of their last migraine attack.
5. Patients who have not taken any acute migraine or pain medication within 48 hours prior to dosing (including OTC products).
6. Patients who have a pain rating of Moderate or Severe (on a None-Mild- Moderate-Severe Scale) prior to dosing.
7. Patients who speak, read, and understand English and are willing and able to provide written informed consent on an IRB approved form prior to the initiation of any study procedures.
8. Patients who are willing and able to comply with the study schedule and requirements, are willing and able to travel to the Clinical Research Unit (CRU) for treatment and stay at the CRU for approximately a 4-6 hour period, and agree to return to the clinic within 5 working days of use of the investigational treatment.
9. Patients who are in good general health prior to study participation as determined by a detailed medical history, physical examination, 12-lead ECG, blood chemistry profile, hematology, urinalysis, and in the opinion of the Principal Investigator.
10. Female participants (if of child-bearing potential and sexually active) and male participants (if sexually active with a partner of child-bearing potential) who agree to use a medically acceptable and effective birth control method throughout the study and for one week following the end of the study. Medically acceptable methods of contraception that may be used by the participant and/or his/her partner include abstinence, birth control pills or patches, diaphragm with spermicide, intrauterine device (IUD), condom with foam or spermicide, vaginal spermicidal suppository, surgical sterilization, and progestin implant or injection. Prohibited methods include: the rhythm method, withdrawal, condoms alone, or diaphragm alone.

Exclusion Criteria:

1. Patients who are currently taking antipsychotics, tricyclic antidepressants, valproate, barbiturates, benzodiazepines, or lithium must be excluded.
2. Patients with a history of contraindications to anticholinergics (bowel obstruction, urinary retention, acute glaucoma) must be excluded.
3. Patients with a history of allergy or intolerance to dibenzoxazepines (loxapine and amoxapine) must be excluded.
4. Patients with a history of extra-pyramidal disorders, movement disorders including Parkinson's disease, and patients with a history of neuroleptic malignant syndrome must be excluded.
5. Female patients who have a positive pregnancy test at screening or during randomization visit, or are breastfeeding must be excluded.
6. Patients who have a history within the past year of drug or alcohol dependence or abuse as defined by DSM-4 must be excluded.
7. Patients who have a history of syncope, unstable angina, myocardial infarction (within 6 months), congestive heart failure, transient ischemic attack, or pheochromocytoma must be excluded.
8. Patients who have a history of a major neurological disorder other than migraine (seizure disorder, subarachnoid bleeding, stroke, brain tumor) must be excluded.
9. Patients who have any other disease(s), by history, physical examination, or laboratory abnormalities (ALT or AST > 2-fold the upper limit of normal, Bilirubin > 1.5 mg/dL, or creatinine > 1.8 mg/dL) or that in the investigator's opinion, would present undue risk to the patient or may confound the interpretation of study results must be excluded.
10. Patients who have a history of asthma or chronic obstructive lung disease should be excluded.
11. Patients who have received an investigational drug within 30 days prior to the Screening Visit must be excluded.
12. Patients who are considered by the investigator, for any reason, to be an unsuitable candidate for receiving loxapine, or unable to use the inhalation device, must be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2007-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Egilius Spierings, MD, Principal Investigator — MedVadis Research Corporation
Locations (1):
- Medvadis, Wellesley Hills, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD submitted to regulatory authorities. Others may contact Alexza Pharmaceuticals, Inc. Please send your request to ClinicalTrialsInfo@alexza.com

RESULTS

PARTICIPANT FLOW:
Groups:
- 1.25 mg Staccato Loxapine: 1.25 mg ADASUVE, single dose
  Staccato Loxapine
- 2.5 mg Staccato Loxapine: 2.5 mg ADASUVE, single dose
  Staccato Loxapine
- 5 mg Staccato Loxapine: 5 mg ADASUVE, single dose
  Staccato Loxapine
Period: Overall Study
Arm/Group | Staccato Placebo | 1.25 mg Staccato Loxapine | 2.5 mg Staccato Loxapine | 5 mg Staccato Loxapine
Started | 39 | 43 | 43 | 43
Completed | 39 | 42 | 43 | 43
Not Completed | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Staccato Placebo | 1.25 mg Staccato Loxapine | 2.5 mg Staccato Loxapine | 5 mg Staccato Loxapine | Total
Number analyzed (Participants) | 39 | 43 | 43 | 43 | 168
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 39 | 43 | 43 | 43 | 168
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (10.94) | 41.7 (13.09) | 38.5 (11.89) | 42.3 (12.68) | 41.1 (2.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 38 | 32 | 35 | 134
  Male | 10 | 5 | 11 | 8 | 34
Region of Enrollment [Number; unit: participants]
  United States | 39 | 43 | 43 | 43 | 168

OUTCOME MEASURES:

1. Primary Outcome: Pain-relief Response (Pain Severity of NONE or MILD) at 2 Hours
Description: The primary efficacy endpoint was Pain-relief response as defined by the International Headache Society (Pain-IHS) as a pain severity of NONE or MILD.
  Intent to treat (ITT) with last observation carried forward (LOCF)
Time Frame: Baseline and 2 h post-dose
Population: ITT Population with LOCF
Measure: Number; unit: participants
Arm/Group | Staccato Placebo | 1.25 mg Staccato Loxapine | 2.5 mg Staccato Loxapine | 5 mg Staccato Loxapine
Number analyzed (Participants) | 39 | 43 | 43 | 43
participants | 20 | 29 | 34 | 33
Statistical Analysis 1: Comparison: Staccato Placebo vs 5 mg Staccato Loxapine; Test type: Superiority; p = 0.0212, Fisher Exact
Statistical Analysis 2: Comparison: Staccato Placebo; Test type: Superiority; p = 0.0106, Fisher Exact

2. Secondary Outcome: Pain-free at 2 Hours
Description: Pain-free (Pain-IHS) at the 2 hour time point
Time Frame: Baseline and 2 h post-dose
Population: ITT with LOCF Population
Measure: Count of Participants; unit: Participants
Arm/Group | Staccato Placebo | 1.25 mg Staccato Loxapine | 2.5 mg Staccato Loxapine | 5 mg Staccato Loxapine
Number analyzed (Participants) | 39 | 43 | 43 | 43
Participants | 3 | 12 | 13 | 9
Statistical Analysis 1: Comparison: Staccato Placebo vs 2.5 mg Staccato Loxapine; Test type: Superiority; p = 0.0123, Fisher Exact
Statistical Analysis 2: Comparison: Staccato Placebo vs 1.25 mg Staccato Loxapine; Test type: Superiority; p = 0.0228, Fisher Exact

3. Other Pre Specified Outcome: Responders, Sustained Freedom From Pain
Description: The percentages of patients with sustained freedom from pain (pain-free at 2 hours after dosing with no rescue medication and no recurrence of headache from 2 to 24 hours)
Time Frame: Baseline through 24 h post-dose
Population: ITT with LOCF Population
Measure: Count of Participants; unit: Participants
Arm/Group | Staccato Placebo | 1.25 mg Staccato Loxapine | 2.5 mg Staccato Loxapine | 5 mg Staccato Loxapine
Number analyzed (Participants) | 39 | 43 | 43 | 43
Participants | 3 | 9 | 11 | 7
Statistical Analysis 1: Comparison: Staccato Placebo vs 2.5 mg Staccato Loxapine; Test type: Superiority; p = 0.0409, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were considered treatment related from the first exposure to study treatment until 30 days after the last treatment
Description: Adverse events (AEs) were assessed at 9 pre-specified time points as well as whenever spontaneously reported by the subjects or study staff
Arm/Group | Staccato Placebo | 1.25 mg Staccato Loxapine | 2.5 mg Staccato Loxapine | 5 mg Staccato Loxapine
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/43 | 0/43 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/43 | 0/43 | 0/43
Other Adverse Events (participants affected / at risk) | 14/39 | 18/43 | 21/43 | 27/43
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Staccato Placebo (N=39) | 1.25 mg Staccato Loxapine (N=43) | 2.5 mg Staccato Loxapine (N=43) | 5 mg Staccato Loxapine (N=43)
Dry Mouth (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Dysgeusia (Gastrointestinal disorders) | 5 (5) | 8 (8) | 10 (10) | 16 (16)
Hypoaesthesia Oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Oral Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Fatigue (General disorders) | 3 (3) | 0 (0) | 3 (3) | 6 (6)
Disturbance in Attention (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
Somnolence (Nervous system disorders) | 5 (5) | 2 (2) | 10 (10) | 10 (10)
Pharyngeal Hypoaesthesia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less